CLINICAL TRIAL: NCT01817088
Title: Sub-thalamic Nucleus Stimulation in Parkinson Disease: Comparison of a Two-steps Electrophysiological Approach Under Local and General Anesthesia and a One-step Approach Under General Anesthesia
Brief Title: Sub-thalamic Nucleus Stimulation in Parkinson Disease
Acronym: PARKEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CHUBX 2012/07
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Parkinson's Disease
Keywords: Deep Brain Stimulation (DBS); Parkinson disease; Stereotaxis Technique; Subthalamic nucleus
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- New targeting procedure without electrophysiology (Experimental): Patients with the high precision procedure under general anesthesia alone without electrophysiological stimulation
  Interventions: Procedure: New targeting procedure without electrophysiology
- Classical neurosurgical procedure (Active Comparator): patients with a first step of electrode implantation under awake surgery with electrophysiological control followed by a second step under general anesthesia
  Interventions: Procedure: Classical neurosurgical procedure

INTERVENTIONS:
Procedure: New targeting procedure without electrophysiology — It is a neurosurgical procedure of electrodes implantation in the sub thalamic nuclei under general anaesthesia using a new targeting procedure without electrophysiology.
  Arms: New targeting procedure without electrophysiology
Procedure: Classical neurosurgical procedure — It is a neurosurgical procedure of electrodes implantation in the sub thalamic nuclei under awake surgery with electrophysiological control. A second surgical step is performed to implant the subcutaneous stimulation device, under general anesthesia.
  Arms: Classical neurosurgical procedure

SUMMARY:
Deep brain stimulation (DBS) is an established procedure for the symptomatic treatment of Parkinson's disease. This procedure performed in two steps using electrophysiology. This study is a prospective, randomized and monocentric study to compare two DBS procedures with or without electrophysiology.

A better control of targeting and trajectory is necessary before not using electrophysiology, which is the reference procedure. A new definition of sub thalamic nuclei with new MRI stereotactic landmarks, the use of surgical robot (Neuromata Renishaw) and the use of operative imaging (O-arm) could allow the implantation of electrode in sub-thalamic nuclei without the need of electrophysiology.

Two groups of patients will be followed: a first group of patients with a procedure under general anesthesia alone without electrophysiological stimulation and a second smaller group of patients with a first step of electrode implantation under awake surgery with electrophysiological stimulation followed by a second step under general anesthesia for the implantation of stimulator.

Clinical results will be assessed at 6 months after implantation.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) is an established procedure for the symptomatic treatment of Parkinson's disease. This procedure performed in two steps using electrophysiology (Limousin et al., 1995) to register the activity of the sub-thalamic nucleus and test the efficacy of stimulation while the patient is awake. A second procedure is needed a few days later to implant the stimulation device under general anaesthesia. The duration of the first procedure is long because of a necessary time of deep stimulation to control the target before definitive implantation. Firstly, the long time of procedure causes pain for the patient. Secondly, the time of procedure, and thus of electrophysiology, is correlated with a rate of device infection of 5 % - 6 % (Hamani et al., 2006; Kenney et al., 2007; Sillay et al., 2008; Doshi et al., 2011). Thirdly, the introduction of several microelectrodes increases the risk of operative and postoperative haemorrhages, estimated at 1 % (Kenney et al., 2007; Sansur et al., 2007; Voges et al., 2007; Bhatia et al., 2008). Moreover, Foltynie et al. (2011) described 12/79 patients treated under general anaesthesia alone with the same post operative results than those who were firstly treated under local anaesthesia.

A better control of targeting and trajectory is necessary before not using electrophysiology, which is the reference procedure. A new definition of sub thalamic nuclei with new MRI stereotactic landmarks, the use of surgical robot (Neuromata Renishaw) and the use of operative imaging (O-arm) could allow the implantation of electrode in sub-thalamic nuclei without the need of electrophysiology. (Caire et al. 2012, In press).

This study is a prospective, randomized and monocentric study. The randomization will be made according to a ratio 2:1 in favour of the technique without electrophysiology. Two groups of patients will be followed: a first group of patients with a procedure under general anesthesia alone without electrophysiological stimulation and a second smaller group of patients with a first step of electrode implantation under awake surgery with electrophysiological stimulation followed by a second step under general anesthesia.

After a preoperative assessment, a end-point evaluation at 6 months after implantation will complete the follow-up.

The stimulation efficacy (UPDRS-3) and the post operative adverse effects will be noticed.

This study will also evaluate the occurrence of a post-traumatic stress disorder (PTSD) in Parkinson disease patients operated under deep brain stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Age : between 18 and 70 years old
* Parkinson disease in fluctuation state despite the use of an optimal medical treatment
* Dopa sensibility higher than 50% with the L-DOPA test
* Normal MRI
* Mattis Scale > 130
* Surgical indication approved by a multidisciplinary team
* Patient covered by a social insurance
* Informed consent signed by patient and investigator

Exclusion Criteria:

* Patients with surgical or anesthetic contraindications
* Cerebral atrophy or signal abnormalities on MRI
* Severe Depressive State : The Beck Scale score > 15
* Women of childbearing potential without efficient contraceptive mean
* Need of long-term antithrombotic treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03-11 (Actual); Primary Completion 2016-09-09 (Actual); Study Completion 2016-09-09 (Actual)

PRIMARY OUTCOMES:
the ratio of preoperative and postoperative UPDRS 3 score | 6 month
  The primary outcome is defined after six months of sub-thalamic nucleus deep brain stimulation with the ratio of preoperative and postoperative UPDRS 3 score. The ratio is : (post operative UPDRS 3 OFF medicine and OFF stimulation- post operative UPDRS 3 OFF medicine ON stimulation)/(post operative UPDRS 3 OFF medicine OFF stimulation)

SECONDARY OUTCOMES:
Stimulation efficacy | 6 month
  Efficacy with the ratio : (Preoperative UPDRS 3 OFF medicine - post operative UPDRS 3 OFF medicine ON stimulation)/( preoperative UPDRS 3 OFF medicine )
The variance of improvement mean for the "high precision" technique | 6 month
  The variance of improvement mean for the "high precision" technique
Percentage of patients with an improvement of UPDRS III score | 6 month
  Percentage of patients with an improvement of UPDRS III score of 35%, 50% et 65%
The Calculated preoperative and post operative (6 months) equivalent dose of L-DOPA and the decrease of between preoperative and post operative period (6 months). | 6 month
  The Calculated preoperative and post operative (6 months) equivalent dose of L-DOPA and the decrease of between preoperative and post operative period (6 months).
Percentage of patients with failure of the new surgical technique defined with an improvement of less than 35 % with the UPDRS 3 score and an electrode located more than 4 mm from the target | 6 month
  Percentage of patients with failure of the new surgical technique defined with an improvement of less than 35 % with the UPDRS 3 score and an electrode located more than 4 mm from the target
Quality of Life | 6 month
  Quality of Life scale : PDQ-39
Non motor items of UPDRS score in the high precision technique under general anesthesia alone | 6 month
  Non motor items of UPDRS score in the high precision technique under general anesthesia alone
Adverse effects and complications | 6 month
  Adverse effects and complications : infection, haemorrhages, paresthesia, hypophonia and dyskinesia
Percentage of improvement in patients with the reference technique | 6 month
  Percentage of improvement in patients with the reference technique (electrophysiological approach in awake surgery)
Compare the technical feasibility for both surgeries based on the number of electrodes implanted in the target | after surgery
  Compare the technical feasibility for both surgeries based on the number of electrodes implanted in the target
Operative and postoperative surgical adverse effects. | 6 month
  Operative and postoperative surgical adverse effects.
Evaluate the influence of two operative procedures on the onset and maintenance of post-operative PTSD | 6 month
  Evaluate the influence of two operative procedures on the onset and maintenance of post-operative PTSD
Evaluate the influence of two operative procedures on the level of preoperative anxiety and the time course of this anxiety | 1, 3 and 6 month
  Evaluate the influence of two operative procedures on the level of preoperative anxiety and the time course of this anxiety
Differentiate thymic and cognitive factors potentially predictors of the occurrence of post-surgical PTSD | 6 month
  Differentiate thymic and cognitive factors potentially predictors of the occurrence of post-surgical PTSD
Evaluate the long-term effects of the two operating procedures on thymic and cognitive state | 6 month
  Evaluate the long-term effects of the two operating procedures on thymic and cognitive state
Evaluate the dose of irradiation received by patients during surgery in both procedures | During surgery

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel CUNY, MD-PhD, Principal Investigator — University Hospital Bordeaux, France; Antoine BENARD, MD, Study Chair — University Hospital Bordeaux, France
Locations (1):
- University Hospital, Bordeaux, France

REFERENCES:
- [Background] Bronstein JM, Tagliati M, Alterman RL, Lozano AM, Volkmann J, Stefani A, Horak FB, Okun MS, Foote KD, Krack P, Pahwa R, Henderson JM, Hariz MI, Bakay RA, Rezai A, Marks WJ Jr, Moro E, Vitek JL, Weaver FM, Gross RE, DeLong MR. Deep brain stimulation for Parkinson disease: an expert consensus and review of key issues. Arch Neurol. 2011 Feb;68(2):165. doi: 10.1001/archneurol.2010.260. Epub 2010 Oct 11. PMID 20937936
- [Background] Cuny E, Guehl D, Burbaud P, Gross C, Dousset V, Rougier A. Lack of agreement between direct magnetic resonance imaging and statistical determination of a subthalamic target: the role of electrophysiological guidance. J Neurosurg. 2002 Sep;97(3):591-7. doi: 10.3171/jns.2002.97.3.0591. PMID 12296643
- [Background] Ferrara J, Diamond A, Hunter C, Davidson A, Almaguer M, Jankovic J. Impact of STN-DBS on life and health satisfaction in patients with Parkinson's disease. J Neurol Neurosurg Psychiatry. 2010 Mar;81(3):315-9. doi: 10.1136/jnnp.2009.184127. Epub 2009 Sep 1. PMID 19726415
- [Background] Kenney C, Simpson R, Hunter C, Ondo W, Almaguer M, Davidson A, Jankovic J. Short-term and long-term safety of deep brain stimulation in the treatment of movement disorders. J Neurosurg. 2007 Apr;106(4):621-5. doi: 10.3171/jns.2007.106.4.621. PMID 17432713
- [Background] Kleiner-Fisman G, Herzog J, Fisman DN, Tamma F, Lyons KE, Pahwa R, Lang AE, Deuschl G. Subthalamic nucleus deep brain stimulation: summary and meta-analysis of outcomes. Mov Disord. 2006 Jun;21 Suppl 14:S290-304. doi: 10.1002/mds.20962. PMID 16892449
- [Background] Limousin P, Krack P, Pollak P, Benazzouz A, Ardouin C, Hoffmann D, Benabid AL. Electrical stimulation of the subthalamic nucleus in advanced Parkinson's disease. N Engl J Med. 1998 Oct 15;339(16):1105-11. doi: 10.1056/NEJM199810153391603. PMID 9770557
- [Background] Maltete D, Navarro S, Welter ML, Roche S, Bonnet AM, Houeto JL, Mesnage V, Pidoux B, Dormont D, Cornu P, Agid Y. Subthalamic stimulation in Parkinson disease: with or without anesthesia? Arch Neurol. 2004 Mar;61(3):390-2. doi: 10.1001/archneur.61.3.390. PMID 15023817
- [Derived] Engelhardt J, Caire F, Damon-Perriere N, Guehl D, Branchard O, Auzou N, Tison F, Meissner WG, Krim E, Bannier S, Benard A, Sitta R, Fontaine D, Hoarau X, Burbaud P, Cuny E. A Phase 2 Randomized Trial of Asleep versus Awake Subthalamic Nucleus Deep Brain Stimulation for Parkinson's Disease. Stereotact Funct Neurosurg. 2021;99(3):230-240. doi: 10.1159/000511424. Epub 2020 Nov 30. PMID 33254172